CLINICAL TRIAL: NCT02706496
Title: Age-related Changes in Posture Control and Cortex Activity Under a Dynamic Perturbation
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014-01-003C
Record Dates: First submitted 2015-08-25; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Aging
Keywords: aging of elderly; falling prevention; electroencephalography; postural control; biomechanics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- young adults (20-35yr): The participants were first screened by the telephone interview, the inclusion criterion contained: able to walk and climb the stairs without assistive devices, could follow the instructions, and without well-known balance related diseases or impairments. With the disease of cardiac and pulmonary system, neuromusculoskeletal system, vision, vestibular apparatus, dizziness experience or cognitive deficit would be excluded the study.
- middle age(45-60yr): The participants were first screened by the telephone interview, the inclusion criterion contained: able to walk and climb the stairs without assistive devices, could follow the instructions, and without well-known balance related diseases or impairments. With the disease of cardiac and pulmonary system, neuromusculoskeletal system, vision, vestibular apparatus, dizziness experience or cognitive deficit would be excluded the study.
- elderly(65-74yr): The participants were first screened by the telephone interview, the inclusion criterion contained: able to walk and climb the stairs without assistive devices, could follow the instructions, and without well-known balance related diseases or impairments. With the disease of cardiac and pulmonary system, neuromusculoskeletal system, vision, vestibular apparatus, dizziness experience or cognitive deficit would be excluded the study.

SUMMARY:
With aging, the elderly decreased ability to control postural balance will be accompanied by increased risk of falling (Berg et al, 1992;. Tinetti et al, 1988). According to previous studies, it showed that the elderly over 65 years fall each year probability was 30 %, and it increased with age (Skelton, & Todd, 2004). In view of this, age-related posture control has become important issues of modern preventive medicine and family care.

DETAILED DESCRIPTION:
Many clinical studies have been developed assessment tools and measurements for clinical staff to provide balanced assessment and intervention. However, the factors of affecting postural control are diverse and complex, not all tools or measurement could effectively detect a risk of falling. In daily living, the postural control involved integration of sensation, biofeedback, movement response, and kinesthetic sense to maintain postural stability, and finally integrated into the neuromuscular system and coordination to help achieve the perfect postural control. Current clinical tools used to assess the fall or research methods to detect the incidence of falls and the lack of effective relevant and contradictory, and it's difficult to effectively evaluate the risk of falls (Gates, et al, 2008).

With the development of postural balance issues associated with aging process in older people, there is no set of standardized equipment, and lack of effective methods for the assessment of normal and older people who fall. In response to these problems, if we can provide a virtual reality interfaces, and with daily living activities as gait, across obstacles activity, sit to stand, will be able to better meet the desire to explore the issue of real significance to enhance researchers for aging, motion analysis, and brain cortex activity mechanism in postural control mechanism.

ELIGIBILITY:
Inclusion Criteria:

* able to walk and climb the stairs without assistive devices,
* could follow the instructions, and
* without well-known balance related diseases or impairments.

Exclusion Criteria:

* With the disease of cardiac and pulmonary system, neuromusculoskeletal system, vision, vestibular apparatus, dizziness experience or cognitive deficit would be excluded the study.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The volunteers from the community will be recruited in this study, the inclusion criterion contained: able to walk and climb the stairs without assistive devices, could follow the instructions, and without well-known balance related diseases or impairments. With the disease of cardiac and pulmonary system, neuromusculoskeletal system, vision, vestibular apparatus, dizziness experience or cognitive deficit would be excluded the study.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
center of pressure | 3 minutes for 20 trial
  0.5m pressure mat (RSscan, Inc., Belgium)

SECONDARY OUTCOMES:
cortex power spectrum density | 3 minutes for 20 trial
  32-channel Ag/AgCl Quick-Cap and NuAmps digital amplifier (Neuroscan, El Paso, TX, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Tsui-Fen Yang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mierau A, Hulsdunker T, Struder HK. Changes in cortical activity associated with adaptive behavior during repeated balance perturbation of unpredictable timing. Front Behav Neurosci. 2015 Oct 14;9:272. doi: 10.3389/fnbeh.2015.00272. eCollection 2015. PMID 26528154